CLINICAL TRIAL: NCT03946813
Title: The Efficacy of Platelets Rich Plasma (PRP) for Ovarian Rejuvenation
Brief Title: The Efficacy of Platelets Rich Plasma for Ovarian Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Kindy College of Medicine (Other)
Collaborators: High Institute for Infertility Diagnosis and Assisted Reproductive Technologies (Unknown)
Responsible Party: Principal Investigator, Yousif Abdulraheem, Professor, Al-Kindy College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12 Al-KindyCM
Record Dates: First submitted 2019-05-06; First posted 2019-05-13 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2019-10

CONDITIONS: Infertility, Female
Keywords: Ovarian Rejuvenation , Infertility
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Poor ovarian reserve (Experimental): Infertile women with poor ovarian reserve
  Interventions: Other: Autologous PRP preparation

INTERVENTIONS:
Other: Autologous PRP preparation — For each patient, autologous PRP preparation havs to be injected to both ovaries and ultrasound (US) guide
  Other Names: Plasma Rich Platelets

SUMMARY:
In recent years, an increased approach has appeared in the use of autologous blood products to assist tissue and organ healing. Application of platelet rich plasma (PRP) has emerged as a potential solution for infertile women with poor ovarian reserve in reproductive specialty.

DETAILED DESCRIPTION:
Quantitative and qualitative functional improvement of ovarian function has been reported in several studies after using autologous PRP in a reproductive field. Ovarian rejuvenation, stimulating the ovaries to produce new eggs after injecting PRP, can offer hope for renewed fertility to women with poor reserve volume, advanced maternal age, or either naturally occurring or premature menopause. But, these encouraging results should be supported by several new studies.

This study aimed to estimate the efficacy of trans-vaginal ovarian injection with PRP in rejuvenates ovaries in woman with poor ovarian reserve, and to assess any association of some women variables (age, menstrual status, parity, BMI) as predicting factors in success of ovarian injection with PRP.

ELIGIBILITY:
Inclusion Criteria:

1. Menopause or peri-menopause under the age of 50.
2. Premature ovarian insufficiency which is ovarian failure before the age of 40.
3. Woman with primary ovarian failure of any cause.

Exclusion Criteria:

1. A previous injection with any medication, plasma, or PRP
2. Invisible or difficult access ovaries.
3. Medical disease or unfit for anesthesia patient.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women
Enrollment: 50 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Follicle-stimulating hormone (FSH) concentration | 4 weeks
  Before after intervention measurement
Anti-Müllerian hormone (AMH) concentration | 4 weeks
  Before after intervention measurement
Antral follicles numbers | 4 weeks
  Before after intervention measurement

CONTACTS AND LOCATIONS:
Overall Officials: Thuraya H Abdulla, Professor, Study Director — Arab Board for Medical Specializations
Locations (1):
- High Institute for Infertility Diagnosis and Assisted Reproductive Technologies, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
All data will be managed confidentially

REFERENCES:
- [Result] A